CLINICAL TRIAL: NCT05743907
Title: A Multicenter, Double-blind, Active-controlled, Randomized, Parallel, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of DA-2811 When Added to Ongoing Metformin Monotherapy in Patients with Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of DA-2811 When Added to Ongoing Metformin Monotherapy in Patients with Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA2811_DM_IV
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-2811 (Experimental): DA-2811 + Forxiga placebo
  Interventions: Drug: DA-2811
- Forxiga (Active Comparator): Forxiga + DA-2811 placebo
  Interventions: Drug: Forxiga

INTERVENTIONS:
Drug: DA-2811 — DA-2811 Group: DA-2811 + Forxiga placebo
  Arms: DA-2811
Drug: Forxiga — Forxiga Group: Forxiga + DA-2811 placebo
  Arms: Forxiga

SUMMARY:
This study is a multicenter, double-blind, active-controlled, randomized, parallel, phase IV clinical trial to evaluate the efficacy and safety of DA-2811 when added to ongoing metformin monotherapy in patients with type 2 diabetes who have inadequate glycemic control

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 7.0%≤HbA1c≤10.0% at screening
* Subjects treated with 1,000mg/day or higher dose of metformin for at least 8 weeks prior to screening
* Subjects with 18.5kg/m2≤BMI≤40kg/m2 at screening
* Subject who is willing and able to provide informed consent indicating that they understand the purpose and procedures required for the study

Exclusion Criteria:

* Subjects with fasting plasma glucose≥240mg/dL at screening
* Patients with type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* Subject with ALT and AST 3 times or higher than upper normal range
* Subject with history of myocardial infarction, cerebral infarction within 3 months prior to screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
HbA1c(%) | Change from baseline at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: Yes